CLINICAL TRIAL: NCT06292143
Title: AI4HOPE - Artificial Intelligence Based Health, Optimism, Purpose, and Endurance in Palliative Care Ofr Dementia: Pilot Study 2 Digital Dementia Care Planning
Brief Title: AI4HOPE Pilot Study 2 Digital Dementia Care Planning
Acronym: AI4HOPE2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bonn (Other)
Collaborators: University College Cork (Other); University of Leeds (Other); Fundacion Intras (Unknown); Universidade do Porto (Other); University Medical Centre Maribor (Other)
Responsible Party: Principal Investigator, Lukas Radbruch, Director Department of Palliative Medicine, University Hospital Bonn, University Hospital, Bonn
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EU101136769-CLIN2
Record Dates: First submitted 2024-02-25; First posted 2024-03-04 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advance Care Planning toolkit (Other): Provision of access to the digital ACP (Advance Care Planning) platform to patients and caregivers, baseline assessment with the ACP digital platform on day 0.
  Information to guide decision making around care and treatment preferences are accessed by patients and carers on days 1 to 7. Where desired, care and treatment preferences are recorded.
  Evaluation of usefulness and burden of the digital platform for ACP on day 7. Content stored on digital platform for ACP shared across care settings to those involved in care of participant on day 8 to 29.
  Evaluation of usefulness and burden of the digital platform for ACP, participant and carer experience of completion. Initial exploration of impact on communication between health and social care professionals, access to timely information to inform clinical decision making, and efficiency savings (e.g. reduction in paper forms and duplication, less time chasing information) on day 90.
  Interventions: Other: Advance Care Planning Toolkit

INTERVENTIONS:
Other: Advance Care Planning Toolkit — Participants or their caregivers will access the digital platform for advance care planning

SUMMARY:
This pilot study will test a digital care planning decision support system for patients with dementia.

DETAILED DESCRIPTION:
The clinical study is part of an EU-funded project on the use of artificial intelligence for patients with dementia. This study will test a digital toolkit for advance care planning and decision making for patients with dementia and pilot-test this digital support system for feasibility and acceptability.

Other workpackages of the AI4HOPE project will design a digital technology platform to provide relevant, timely and appropriate information for people with dementia and their carers, and to facilitate them to document their goals, wishes, and preferences for future care.

Patients with mild to moderate dementia will be recruited for the pilot study in the six participating countries. The study population includes all types of dementia without stratification, as the aim of the study is to develop a digital technology platform to facilitate ACP for clinical practice in any patient with cognitive impairment from any type of dementia.

Even though the digital platform could be adapted to be useful for patients with advanced dementia and more severe cognitive impairment, or for use just by their families, the pilot study will recruit only patients with mild or moderate dementia, who will still be able to provide informed consent, and who will be able to self-assess for patient-related outcome or patient-related experience measures to inform the assessment of the digital technology platform.

Patients with dementia treated in the participating study centers will be screened for inclusion criteria and, if suitable will be invited to participate. The study will be performed for up to 90 days, with optional extension to 180 days according to patients' preferences.

Patients with baseline data and at least one interaction with the digital platform and data completed before and after that interaction will be included in the evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Mild or moderate dementia of any type
* Montreal Cognitive Assessment (MoCA) score of 16-25
* Living at home, or in residential or nursing home care
* Receiving adequate social support

Exclusion Criteria:

* Moderate/severe cognitive impairment (MoCA < 16)
* No cognitive impairment (MoCA >25)
* Inpatient or acute hospital treatment
* Infectious diseases or lokal skin conditions preventing the use of wearable body sensors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of digital ACP-platform, the Dementia Journey Companion (DJC) | 30 days
  Participant feedback on feasibility, usefulness and burden of ACP-platform; acceptability of content included in the ACP-platform for participantd, user satisfaction with conversational support and suc-cess rate in achieving communicative goals, answering questions and providing guidance.

SECONDARY OUTCOMES:
Effect of DJC on documentation of ACP | 30 days
  Rating of benefit by health care professionals.
Completion rate of preference documentation | 30 days
  Completion rate of preference documentation across domains (daily living, medical, end-of-life) and frequency of use; frequency of chatbot interactions; number of memories, stories, and preferences documented.
Assessment of pain, distress and anxiety | 30 days
  Assessment of pain, distress and anxiety (PROM as part of assessment toolkit).

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Radbruch, MD, Principal Investigator — Department of Palliative Medicine, University Hospital Bonn

IPD SHARING:
Plan to Share IPD: No